CLINICAL TRIAL: NCT05643391
Title: RadioEmbolizaTion Using hOlmium-166 in Patients With Unresectable Hepatocellular Carcinoma: Prospective, Open Label, Single-center Pilot Study
Brief Title: Safety and Feasibility of Radioembolization Using Ho-166 in Patients With Unresectable Hepatocellular Carcinoma
Acronym: RETOUCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2020/226
Record Dates: First submitted 2022-11-07; First posted 2022-12-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radioembolization; Holmium-166; Transarterial locoregional therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): The treatment will include 1 preparatory angiography followed by treatment at a maximum 2 weeks interval. Dosimetry MRI will be performed just before and immediately after treatment. SPECT CT will be performed three days after treatment.
  The activity of 166Ho that must be administered to a patient will depend on the tumor perfusion and absorbed dose linked to this activity.Q-SuiteTM 2.0 will be used, more precisely a dosimetry software to perform an optimal compartmental predictive dosimetry:
  - minimum 150 Gy to the tumor, maximum 60 Gy to non-tumoral liver, maximum 30 Gy lung shunt fraction.
  Interventions: Radiation: Radioembolization using Holmium-166

INTERVENTIONS:
Radiation: Radioembolization using Holmium-166 — This technic consists of the intra-arterial infusion of smaller beads that are loaded with a radioactive isotope (yttrium-90), and it relies on the beta radiation emitted by the isotope to induce tumor necrosis, with a minor contribution from microembolization and without risk of ischemia of the remaining liver.

SUMMARY:
Background: Hepatocellular carcinoma (HCC) accounts for 90% of primary liver cancers and represents a growing health problem worldwide. Most patients present locally advanced disease and are candidates for palliative transarterial locoregional treatment. Transarterial radioembolization (TARE) using 90Y has been used for more than a decade for patients with advanced disease. The use of 166Ho could offer a more personalized approach in terms of imaging and dosimetry. Aim: to evaluate the feasibility and safety of TARE using 166Ho in a selected population of HCC patients and assess the biological peripheral response to this therapy. Materials and methods: In this open-label, prospective, non-randomized, singlecenter pilot study, 20 patients with unresectable hepatocellular carcinoma will undergo TARE using 166Ho. The primary outcome is the feasibility of 166Ho radioembolization as well as the assessment of safety and toxicity profiles (CTAE V5.0). Secondary outcomes include the evaluation of efficacy of 166Ho radioembolization in unresectable hepatocellular carcinoma, according to mRECIST and metabolic criteria, as well as the impact on the tumor marker alpha-fetoprotein (AFP), assessment of biodistribution/dosimetry using a "scout dose" and time to progression (TTP). A substudy will assess the hepatic function using 99mTc-IDA hepato-biliary scintigraphy (HBS) and the comparison between "pre-scout" HBS and HBS just after "scout dose". Finally, blood samples will be collected at different time points in order to explore the biological peripheral response to these therapies. Perspectives: The newly developed 166Ho-microspheres have distinctive advantages over the existing 90Ymicrospheres with improved dosimetry that represents a prerequisite for optimal safety and efficacy.

DETAILED DESCRIPTION:
Primary liver cancer is a growing health problem worldwide. Hepatocellular carcinoma (HCC) represents more than 90% of primary liver cancers and is considered to be the fifth most common cancer and the second leading cause of cancer-related deaths, with the majority being associated to cirrhosis.

Choosing the most suitable treatment option depends not only on the tumor stage, but also on the severity of the underlying liver disease and performance status. Current guidelines consider the Barcelona Clinic Liver Cancer (BCLC) staging system as the algorithm of choice for tumor staging and therapeutic options, taking into account tumor burden, Child-Pugh class and performance status (ECOG).

Surgical approach, such as resection and liver transplantation, and radiofrequency (RFA) represent the curative treatment options. Despite screening of at-risk populations, most patients are diagnosed with locally advanced disease (BCLC B - intermediate stage) and will not be suitable for curative therapies. Moreover, only HCC within the "Milan" criteria (one nodule < 5 cm or up to three nodules < 3 cm in diameter, without macroscopic vascular invasion or extrahepatic disease) are potential candidates for transplantation. Resection can be proposed only in case of compensated cirrhosis in the absence of portal hypertension and RFA is only possible for small lesions (< 5 cm, < 3 cm in diameter).

Locally advanced HCC is suitable for transarterial locoregional therapies, conducted mostly in a palliative setting. They take advantage on the double vascularization of the liver, with 75% of the parenchymas blood supply coming from the portal vein, while tumor nodules blood supply being almost exclusively provided by the hepatic artery. When macrovascular involvement or extrahepatic disease are discovered, but patients present a good performance status and a compensated liver function (BCLC C), systemic therapy with the tyrosine kinase inhibitor Sorafenib leads to a limited survival benefit, approximately 3 months advantage compared to placebo.

Transarterial chemoembolization (TACE), either conventional (cTACE) or using drug-eluting embolic (DEE) agents, is recommended for patients with BCLC stage B and as "bridging" therapy for liver transplantation candidates while on the waiting list. Furthermore, it has been shown that in selected patients, it can be successfully used as a downstaging treatment to transplantation criteria.

Technically, TACE involves the injection of a chemotherapeutic agent (i.e. doxorubicin), mixed with an embolic material, administered selectively into the feeding arteries of the tumor resulting in tumoral necrosis induced by ischemia and cytotoxic effect.

During the last decade, transarterial radioembolization (TARE) with yttrium-90 microspheres [Y90] was introduced in case of TACE failure or for patients who were not suitable for TACE (i.e.: large tumors or macrovascular invasion). This technic consists of the intra-arterial infusion of smaller beads that are loaded with a radioactive isotope (yttrium-90), and it relies on the beta radiation emitted by the isotope to induce tumor necrosis, with a minor contribution from microembolization and without risk of ischemia of the remaining liver. Its efficacy was reported in several large patient series. Two products are commercially available for TARE. 90Y-labelled resin microspheres (SIR-Spheres; Sirtex Medical, Sydney) and 90Y glass microspheres (TheraSphere; Boston International).

The radioembolization procedure are performed over two different sessions: work-up session and treatment session.

The work-up evaluation starts with an angiography in order to obtain a precise map of the patients' abdominal vascular anatomy and coil embolization might be performed if gastro-intestinal branches arising from the hepatic arteries are found. This will prevent radioactive microspheres, administered into the hepatic artery, from ending up in extrahepatic organs via this route.

The second step of the work-up implies the injection of 150 MBq Technetium-99 m-labeled macro aggregated albumin (99mTc-MAA) in order to predict the distribution pattern of 90Y-microspheres. The uptake of 99mTc-MAA will be visualized by whole body planar imaging and single-photon emission computed tomography (SPECT-CT), including low dose computer tomography of the abdomen. 99mTc-MAA lung shunt fraction will be calculated and lung dosage must not exceed 30 Gy in a single treatment.

In case on an unfavorable 99mTc-MAA workup, the procedure will be repeated, if possible, to detect the cause of the extrahepatic deposition (for example, previously undetected patent extrahepatic vessels arising from the hepatic artery) and a solution will be searched for (for example, more selective placement of the catheter during injection to improve the targeting of the lesion). In the unlikely event no solution can be found and 90Y TARE cannot be performed, the patient will be treated according to best medical practice.

If the work-up will have a favorable outcome, the patients will be re-admitted for the treatment within 15 days.

Several retrospective studies and non-controlled prospective studies have shown higher rates of objective tumor responses, prolonged time to progression and overall survival for TARE, with study advocating it more effective than TACE as a downstaging tool to curative treatment. Nevertheless its place in the treatment of HCC is still to be defined, especially due to the non-compartmental predictive dosimetry usually performed in recent studies.

Post-treatment calculation of the radiation absorbed dose in the tumors and the healthy liver tissue cannot be easily performed because quantitative PET imaging of the beta-emitting 90Y-microspheres is challenging. New generation microspheres may help to achieve post-treatment dosimetry easily.

New Holmium-166 (166Ho) loaded poly(L-lactic acid) microspheres have been developed at the Department on Radiology and Nuclear Medicine of the University Medical center (UMC) Utrecht and are commercialized by Terumo Europe (QuiremSpheres®). Just like 90Y, 166Ho relies on the emitted beta radiation to induce tumor necrosis. The advantage provided by this isotope is its gamma radiation emission, which allows for quantitative SPECT imaging (166Ho: T1/2 of 27 hours, gamma-radiation 81 keV, beta-radiation 1.8 MeV) and the assessment of the radiation absorbed dose delivered in both the tumor(s) and the remaining part of the liver (i.e. dosimetry). Besides, holmium is a highly paramagnetic metal, and as such may be visualized by MRI. This is useful because quantitative analysis of the MRI scans is possible, including R2* relaxometry for microsphere concentration, and especially useful for medium- and long-term monitoring of the intra-hepatic behavior of the microspheres.

TARE using 166Ho -microspheres underwent a first evaluation in a clinical phase I safety study with an administration system specifically designed for 166Ho radioembolization (HEPAR I, METC 08-450). Fifteen patients with unresectable, chemorefractory liver metastases were enrolled, using a standard dose escalation protocol. They were treated in cohorts of 3 (target absorbed dose 20 Gy, 40 Gy, 60 Gy and 80 Gy). The maximum tolerable radiation dose was 60 Gy. In the 80 Gy cohort, dose-limiting toxicity occurred in two patients: grade four thrombocytopenia, grade three leukopenia, and grade three hypoalbuminaemia in one patient, and grade three abdominal pain in another patient. The most frequently encountered laboratory toxicities (including grade one) were lymphocytopenia, hypoalbuminaemia, raised alkaline phosphatase, raised aspartate aminotransferase, and raised gamma-glutamyltransferase, which were all noted in 12 of 15 patients (80%). Stable disease or partial response regarding target lesions was achieved in 14 of 15 patients (93%, 95% CI 70-99) at 6 weeks and 9 of 14 patients (64%, 95% CI 39-84) at 3 months after TARE. It was concluded that 166Ho radioembolization is feasible and safe for the treatment of patients with unresectable and chemorefractory liver metastases and enables image-guided treatment.

This was followed by a non-randomized single-arm phase II study that included 56 patients with unresectable, chemorefractory liver metastases (HEPAR II METC 11-538). 166Ho radioembolization was performed with a mean liver absorbed dose of 60 Gy. The primary outcome was tumor response of two target lesions on triphasic liver CT scans, 3 months after therapy using modified RECIST criteria as evaluated by three blinded readers. After treatment of 38 eligible patients, the target lesions showed disease control in 73% after 3 months (95% confidence interval [CI], 57 to 85%). The median overall survival was 15.3 months (95% CI, 9.1 to ∞ months). Grade three or four toxic events (according to CTCAE version 4.03 criteria) after treatment included abdominal pain (in 18% of patients), nausea (9%), ascites (3%), gastric stenosis (3%), liver abscesses (3%), paroxysmal atrial tachycardia (3%), REILD (3%), thoracic pain (3%), upper gastrointestinal hemorrhage (3%), and vomiting (3%). Laboratory examination after treatment showed grade three or four toxicities in alkaline phosphatase (70%), γGT (78%), lymphocytes (11%), and ALAT (4%). From the results of this study it was concluded that 166Ho radioembolization induced a favorable tumor response with an acceptable toxicity profile in patients with liver metastases.

The University Medical center (UMC) of Utrecht is currently conducting a third study for patients with HCC (HEPAR Primary, NCT03379844). The primary objective is to evaluate safety and toxicity profile of 166Ho-TARE. HCC patients were not included in previous studies, because underlying liver disease in HCC patients puts a higher demand on safety issues, which should be studied separately.

The investigators aim to evaluate the efficacy and safety of TARE using the newly developed 166Ho-microspheres in our HCC population, at ERASME Hospital. Using 166Ho has distinctive advantages over the existing 90Y-microspheres, making quantitative individualized dose planning possible by means of SPECT and MRI. Accurate dosimetry in radiation treatment is a prerequisite for optimal safety and efficacy evaluation. This is particularly relevant in patients with hepatocellular carcinoma and underlying chronic liver disease, which limits the maximum tolerated absorbed dose that can be applied to the liver.

Regarding this underlying chronic liver disease, assessment of hepatic function with 99mTc-IDA hepatobiliary scintigraphy is routinely performed at Erasme hospital before TARE. However, in classical 90Y TARE workflow, because both MAA and IDA are labeled with 99mTc the predictive dosimetry and the evaluation of the hepatic function with IDA cannot be performed on the same day. The management of the patient and the planning of TARE may be greatly optimized if both predictive dosimetry and evaluation of hepatic function can be performed on the same day. And it becomes possible with the use of 166Ho.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given written informed consent
* Adults ≥ 18 years-old
* Typical imaging or biopsy proven HCC according to EASL-EORTC guidelines (1)
* Unresectable disease, BCLC B, or contraindicated for ablation, resection or transplantation, BCLC A, or BCLC C patients with no extra-hepatic extension, patients on the waiting list for resection or transplantation.
* At least one measurable lesion on multiphasic CT or MRI
* Preserved liver function with Child- Pugh score≤ B7
* ECOG performance status ≤ 1 (Table 2)
* Life expectancy ≥3 months
* Efficient contraception for women
* Platelets ≥ 50000/m3 and PT≥ 50%
* Hemoglobin ≥8.5 g/dl
* Bilirubin ≤ 2 mg/dl
* ASAT/ALAT levels ≤ 5x upper normal limit
* Creatinine ≤ 1.5x upper normal limit

Exclusion Criteria:

* Before work-up:

  * History of progressive, uncontrolled cancer other than HCC presenting liver metastasis.
  * >50% of liver involvement
  * Portal vein thrombosis of the main branch diagnosed on contrast enhanced images. Involvement of the right or left portal main branches and more distal is accepted
  * Evidence of extrahepatic disease
  * Unmanageable intolerance to contrast medium
  * Contraindication to hepatic angiography
  * Digestive hemorrhage due to portal hypertension in the 30 days preceding treatment
  * Previous systemic treatment, radiation therapy, transarterial loco-regional therapy or ablation therapy for HCC
  * Active infection or untreated active hepatitis (if detectable viral HBV load, treatment with a nucleoside analog should be instituted).
  * Pregnancy or breast feeding
  * Ascitis
  * Transjugular intrahepatic portosystemic shunt (TIPS) or portacaval shunt
  * Major surgery withing 4 weeks or incompletely healed surgical incision before starting study therapy
  * Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or severe depression.
  * Patients who are declared incapacitated
* After work-up:

  * Lung absorbed dose > 30 Gy, as calculated using the 166Ho scout dose or 99mTc MAA
  * Uncorrectable extrahepatic deposition of the scout dose activity. Activity in the falciform ligament, portal lymph nodes and gallbladder is accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Achievement of the selective radioembolization with Holmium-166 treatment in patients with HCC | immediately after the SIRT session
  Feasibility will be measured by the number of completed treatments and the percentage of injected activity compared to simulation
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | Day 1
  % of patients with change in clinical, biological and radiological parameters
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | 1 month
  % of patients with change in clinical, biological and radiological parameters
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | 3 months
  % of patients with change in clinical, biological and radiological parameters
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | 6 months
  % of patients with change in clinical, biological and radiological parameters

SECONDARY OUTCOMES:
Evaluation of efficacy of 166Ho radioembolization in unresectable hepatocellular carcinoma, according to mRECIST | 3 months
  mRECIST for HCC lesions: Evaluation of target lesions
  * Complete Response (CR): Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the target lesions
  * Progressive Disease (PD): At least a 20% increase in the sum of the target lesions
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD Evaluation of non-target lesions
  * Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level
  * Incomplete Response/ Stable Disease (SD): Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits
  * Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Evaluation of biodistribution/dosimetry using a scout dose | Day 5
  Tumoral and non-tumoral dose distribution in the liver and dose distribution in the lungs.
Evaluation of tumor response marker alpha-fetoprotein | Baseline,1,3,6 Months
Time to progression (TTP) | 6 months
  Time elapsed from enrolment until objective tumor progression; does not include deaths
Microsphere concentration derived from 1.5T MRI R2* relaxivity measurements | Baseline and immediately after the intervention
Evaluation of efficacy of 166Ho radioembolization in unresectable hepatocellular using metabolic assessments (FDG and choline PET/CT) | 3 months
  % of patients that showed a complete metabolic response (CMR), partial metabolic response (PMR), no metabolic response (SMR), or progressive disease with new lesions.

OTHER OUTCOMES:
Assess the peripheral response to TA-LRT (i.e.: serum levels of tumor necrosis factor (TNF-alfa), interleukine-6 and 8 (IL6, IL8) and vascular endothelial growth factor (VEGF) at different time points of the study) | Baseline, day 1, day 14 and one month
Evaluation of hepatic function using 99mTc-IDA hepato-biliary scintigraphy (HBS) | 3 months
Comparison between "pre-scout" HBS and HBS just after "scout dose" | Baseline and immediately after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gontran VERSET, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Hôpital Universitaire Erasme, ULB, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No